CLINICAL TRIAL: NCT03508401
Title: Transthoracic Echocardiographic Assessment of the Superior Vena Cava Flow Respiratory Variation in ICU Intubated Patients
Brief Title: Transthoracic Echocardiography of the Superior Vena Cava in Intensive Care Units (ICU) Intubated Patients
Acronym: CAVSUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0549
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Intubated Patients; Admission in Intensive Care Unit
Keywords: superior vena cava

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICU intubated patients (Experimental): After inclusion, Echo-Doppler measurements are performed with Vivid S6 model (GE Healthcare France, Lyon, France). The left ventricular outflow tract velocity time index (LVOT TVI) will be measured with this device. Then, a passive leg raising (PLR) will be performed and finally LVOT VTI will be measured again after PLR
  Patients will be classified in two groups according to the hemodynamic response to PLR :
  * Patients are responders if LVOT VTI increases of at least 10% after PLR
  * patients are non-responders if LVOT VTI does not increase or increase of less than 10% after PLR.
  Interventions: Other: Passive leg raising (PLR); Device: Echo-Doppler measurements

INTERVENTIONS:
Other: Passive leg raising (PLR) — PLR is a test that predicts whether cardiac output will increase with volume expansion. By transferring a volume of around 300 mL of venous blood from the lower body toward the right heart, PLR mimics a fluid challenge. However, no fluid is infused and the hemodynamic effects are rapidly reversible, thereby avoiding the risks of fluid overload.
  PLR starts from the semi-recumbent and not the supine position. PLR is performed by adjusting the bed and not by manually raising the patient's legs
Device: Echo-Doppler measurements — Echo-Doppler measurements are performed with Vivid S6 model (GE Healthcare France, Lyon, France). All measurements are recorded at the end of expiration. Echo-Doppler measurements are performed in the upper part of the SVC, approximately 1 to 2 cm below the brachiocephalic vein. From this view, pulse Doppler is performed. Pulse Doppler waves obtained in the SVC are used to obtain velocity time integrals (VTI). Expiratory VTI is named VTImax and inspiratory VTI is named VTImin. These values will allow the calculation of Respiratory variations of the superior vena cava flow (ΔSVCf).
  ΔSVCf is calculated as (VTImax- VTImin )/(1/2(VTImax+ VTImin)).

SUMMARY:
Acute circulatory failure is frequent, affecting up to one-third of patients admitted to intensive care units (ICU). Monitoring hemodynamics and cardiac function is therefore a major concern. Analysis of respiratory diameter variations of the superior vena cava (SVC) is easily obtained with transesophageal echocardiography (TEE) and is helpful to assess fluid responsiveness.

Transthoracic echocardiography (TTE) exploration of the SVC is not used in routine. Recently, micro-convex ultrasound transducers have been marketed and these may be of use for non-invasive SVC flow examination. However, analysis of diameter variations of the SVC with TTE does not seem to be possible since the approach from the supraclavicular fossa does not allow for a good visualization of the SVC walls.

It was recently demonstrated in a short pilot study that TTE examination of the SVC flow with a micro-convex ultrasound transducer (GE 8C-RS) seems both easy to learn and to use (feasibility = 84.9%), and is reproducible in most ventilated ICU patients with an intraclass correlation coefficient for the systolic fraction of the superior vena cava flow of 0.90 (95% confidence interval [0.86-0.93]).

The hypothesis is that cardio-respiratory interactions in intubated-ventilated patients are responsible of SVC flow variations and that the analysis of the SVC flow respiratory variations could be a new predictive tool of fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Admission in ICU after tracheal intubation or tracheal intubation during the ICU stay
* Volume-controlled ventilation with a tidal volume of 8 mL/kg
* Patient or family agreement for the inclusion

Exclusion Criteria:

* Persistence of spontaneous breathing
* Cardiac arrhythmia
* Severe Acute Respiratory Distress Syndrome, defined as PaO2/FIO2 ratio < 100
* Acute right ventricular failure defined by S'VD < 10 cm or Tricuspid Annular Plane Systolic Excursion (TAPSE) < 10 mm measured with Transthoracic Echocardiography (TTE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-05-25 (Estimated); Study Completion 2020-05-25 (Estimated)

PRIMARY OUTCOMES:
ventricular outflow tract velocity time index (LVOT TVI) | The day of inclusion
  Echo-Doppler measurements are performed with Vivid S6 model (GE Healthcare France, Lyon, France). All measurements are recorded at the end of expiration. Echo-Doppler measurements are performed in the upper part of the SVC, approximately 1 to 2 cm below the brachiocephalic vein. From this view, pulse Doppler is performed. Pulse Doppler waves obtained in the SVC are used to obtain velocity time integrals (VTI). Expiratory VTI is named VTImax and inspiratory VTI is named VTImin. These values will allow the calculation of Respiratory variations of the superior vena cava flow (ΔSVCf).
  ΔSVCf is calculated as(VTImax- VTImin )/(1/2(VTImax+ VTImin))

SECONDARY OUTCOMES:
optimal cut-off value of ΔSVCf to predict fluid-responsiveness | The day of inclusion
proportion of patients in which measurement of ΔSVCf is not possible | The day of inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'Anesthésie-Réanimation, Hôpital Edouard Herriot,, Lyon, France